CLINICAL TRIAL: NCT06444737
Title: Contribution of Ondansetron to Preventing Post-Dural Puncture Headaches Following Spinal Anesthesia for Cesarean Sections : A Randomized Controlled Trial
Brief Title: Contribution of Ondansetron to Preventing Post-Dural Puncture Headaches Following Spinal Anesthesia
Acronym: OPDPH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mongi Slim Hospital (Other)
Responsible Party: Principal Investigator, Mhamed Sami Mebazaa, Professor head of anesthesiology and ICU department, Mongi Slim Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ondansetron effect on PDPH
Record Dates: First submitted 2024-05-13; First posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-05

CONDITIONS: Post-Dural Puncture Headache
MeSH Terms: conditions — Post-Dural Puncture Headache | interventions — Ondansetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group O (Experimental): Group ondansetron : parturients receiving intravenous (IV) ondansetron 0.10 mg/ kg diluted in 5 ml normal saline, 5 min before spinal anesthesia
  Interventions: Drug: Intravenous ondansetron
- Group C (Placebo Comparator): Group control : receiving IV normal saline 5 ml (control group) 5 min before spinal anesthesia
  Interventions: Drug: Intravenous normal saline

INTERVENTIONS:
Drug: Intravenous ondansetron — Intravenous (IV) ondansetron 0.10 mg/ kg diluted in 5 ml normal saline, 5 min before spinal anesthesia
  Other Names: ondansetron
  Arms: Group O
Drug: Intravenous normal saline — Intravenous normal saline 5 ml (control group) 5 min before spinal anesthesia
  Other Names: Placebo
  Arms: Group C

SUMMARY:
A prospective, bicentric, randomized, double-blind controlled study including parturients scheduled for elective caesarean delivery under spinal anaesthesia and randomized and assigned to one of the two groups:

Group O ondansetron : receiving Intravenous (IV) ondansetron 0.10 mg/ kg diluted in 5 ml normal saline, 5 min before spinal anesthesia Group C control : receiving IV normal saline 5 ml (control group) 5 min before spinal anesthesia

OBJECTIVE :

To evaluate the efficacy of ondansetron in preventing post-dural puncture headache after spinal anaesthesia for caesarean section.

DETAILED DESCRIPTION:
Spinal anesthesia is the most common anesthetic technique used for Caesarean sections. However, it is not denied from complications.

Post-dural puncture headache is a major complication of spinal anesthesia, with an incidence ranging from 1.5% to 36%.

OBJECTIVE :

To evaluate the efficacy of ondansetron in preventing post-dural puncture headache after spinal anaesthesia for caesarean section.

the investigators conducted a prospective, bicentric, randomized, double-blind controlled study over a period of 07 months from November 2023 to june 2024.

the investigators included in the study all parturients:

* Aged between 18-45 years
* ASA 2
* Between 37 and 41 weeks of gestation
* scheduled for elective caesarean delivery under spinal anaesthesia
* To be delivered by unscheduled caesarean section whose indication does not involve a vital maternal or fetal emergency, according to the Lucas' classification.

The eligible parturients were randomly assigned to two groups through block randomization using computerized random numbers.

were assigned to one of the two parallel groups to receive either :

* Intravenous (IV) ondansetron 0.10 mg/ kg diluted in 5 ml normal saline, 5 min before spinal anesthesia : Group O (Ondansetron)
* Or IV normal saline 5 ml (control group) 5 min before spinal anesthesia : Group C (control)

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-45 years
* ASA 2
* Between 37 and 41 weeks of gestation
* scheduled for elective caesarean delivery under spinal anaesthesia
* To be delivered by unscheduled caesarean section whose indication does not involve a vital maternal or fetal emergency, according to the Lucas' classification

Exclusion Criteria:

* All patients who required :
* more than two attempts for spinal anaesthesia
* conversion to general anesthesia following failure of spinal anesthesia (defined as a sensory block level <T6) or an intraoperative complication (such as hemorrhage or anaphylactic shock).

As well as patients who have subsequently withdrawn their consent for participating to our study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — parturients scheduled for elective caesarean delivery under spinal anaesthesia
Enrollment: 300 (Estimated)
Dates: Start 2023-11-30 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of post-dural punction headache (PDPH) during the first seven postoperative days. | 7 days
  the occurrence of positional headaches at any time postoperatively

SECONDARY OUTCOMES:
day of PDPH's occurence | 7 days
  on postoperatively
day of PDPH's resolution | 7 days
  on postoperatively
Headache severity | 7 days
  assessed by the numerical pain scale from 0 to 10 (0 being no pain and 10 being the maximum unimaginable pain).
Need for analgesic treatment due to headaches | 7 days
  paracetamol or NSAIDs
Occurrence of post-operative nausea and/or vomiting | 7 days
  need of treatement
Mean arterial pressure in mmgh | 3 days
  Mean arterial pressure during hospitalization
heart rate | 3 days
  Mean arterial pressure during hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- Mongi slim hospital, Tunis, Tunisia